CLINICAL TRIAL: NCT04732442
Title: Changes in Inflammatory Response After Immunonutrition Compared to Standard Nutritional Support in Colorectal Cancer Tissue - Randomized Controlled Trial
Brief Title: Changes in Inflammatory Response After Immunonutrition Compared to Standard Nutrition in Colorectal Cancer Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, Prof., MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JagiellonianU-07
Record Dates: First submitted 2021-01-19; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Colon Cancer; Nutrition Aspect of Cancer
Keywords: immunonutrition; colon cancer; inflammatory response; perioperative care; randomized controlled trial
MeSH Terms: conditions — Colonic Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: Randomized 2-arm controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immuno-group (Experimental): The immuno-group will consist of patients who, as part of preoperative nutritional support, used immunonutrition ONS (2x Impact Oral® Nestle, Switzerland per day) for 2 weeks before surgery.
  Interventions: Dietary Supplement: Immunonutrition
- Control-group (Sham Comparator): The control group will consist of patients who, as part of preoperative nutritional support, used standard ONS (3x Fortimel Compact Protein® Nutricia, United Kingdom per day) for 2 weeks before surgery.
  Interventions: Dietary Supplement: Standard Oral Nutritional Support

INTERVENTIONS:
Dietary Supplement: Immunonutrition — Impact Oral® Nestle, Switzerland
  Other Names: Immunonutrition Oral Nutritional Support
  Arms: Immuno-group
Dietary Supplement: Standard Oral Nutritional Support — Fortimel Compact Protein® Nutricia, United Kingdom
  Arms: Control-group

SUMMARY:
It is Randomized Controlled Trial, in which investigators will estimate the impact of the use of immunonutrition support compared to standard nutritional support in the preoperative period in patients with colorectal cancer.

DETAILED DESCRIPTION:
The first choice of treatment in colorectal cancer is surgery. Nutritional support in form of oral nutritional supplements (ONS) in the preoperative period is widely accepted in reducing the incidence of perioperative complications and immunonutrition is generally recommended. However, there is little clinical data regarding the impact of such treatment on a tumor biology.

Investigators want to perform Randomized Controlled Trial to explore the impact of the use of immunonutrition in relation to standard nutritional support in the preoperative period on alternating the expression of inflammatory response cytokines expression and leukocytes infiltration in tumor tissue in patients operated for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colon cancer during preoperative colonoscopy confirmed by histopathological examination.

Exclusion Criteria:

* emergency/urgent operation
* active infection
* inflammatory bowel diseases in history
* other systemic immune disorders
* the necessity of preoperative neoadjuvant treatment (radiotherapy or chemotherapy)
* metastatic disease, or local infiltration of cancer which was described as T4 stage in preoperative CT scan
* patients who were not able to intake at least 85% of administrated ONS doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change in expression of inflammatory cytokines in tumor tissue samples obtained prior and after intervention. | up to 13 months
  Expression of following inflammatory cytokines will be measured: Tumor necrosis factor (TNF-α), Interleukin 8 or chemokine (C-X-C motif) ligand (CXCL8), stromal cell-derived factor 1 (SDF-1a), Chemokine (C-X-C motif) ligand 6 (CXCL6), Chemokine (C-X-C motif) ligand 2 (CXCL2), myeloperoxidase (MPO), Chemokine (C-X-C motif) ligand 1 (CXCL1) prior and after intervention. Measurements of cytokines' tissue concentration will be presented in pg/100ug of total protein.

SECONDARY OUTCOMES:
Changes in tissue neutrophil infiltration after preoperative nutritional intervention in tumor tissue samples obtained prior and after intervention. | up to 13 months
  Neutrophil infiltration will be assessed by counting the number of neutrophils per 10 large microscopic fields.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Pędziwiatr, Prof., Principal Investigator — Jagiellonian University
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No